CLINICAL TRIAL: NCT01449474
Title: Accuracy of MRI-based Patients Matched Instruments and Jig-based Instruments in Total Knee Arthroplasty
Brief Title: Accuracy of MRI-based Patients Matched Instruments vs Jig-based Instruments in Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si050/2554(EC2)
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Patient matched instruments
  Interventions: Device: Patient matched instruments
- Group 2 (Experimental): Jig based instruments
  Interventions: Device: Jig based instruments

INTERVENTIONS:
Device: Patient matched instruments — The patients undergo TKA with using patient matched instruments
  Other Names: The Zimmer Patient Specific Instruments System
  Arms: Group 1
Device: Jig based instruments — The patients undergo TKA with using jig based instruments
  Other Names: Zimmer Nexgen LPS MIS system
  Arms: Group 2

SUMMARY:
Total knee arthroplasty (TKA) is the common and effective procedure for treatment of end-staged knee osteoarthritis. Postoperative alignment of TKA is one of the important factors which effects on survival of prosthesis. High percentage of misalignment has been reported in conventional technique with using the jig based instruments. Several methods and devices were established to solve this problem. Customized or patient matched instruments were the novel technology that made from magnetic resonance imaging (MRI) of lower limb. With using special software to calculate the alignment axis, it was thought that accurate alignment can be achieved by using this instruments. Therefore, the study aimed to compare the accuracy of MRI based patient matched instruments and jig based instruments in TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed primary osteoarthritis of knee and planned to undergo total knee arthroplasty

Exclusion Criteria:

* Previous complex surgery of the affected knee
* Metalic implant in the affected lower limb
* Patients who unable or contraindicated to perform MRI
* Extra-articular deformities of the affected lower limb
* Extensive bone loss of distal femur or/and proximal tibia
* More than 30 degrees of knee flexion contracture
* Unable to perform TKA within 12 weeks after MRI

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The alignment of mechanical axis after TKA | Within 1 month after operation

SECONDARY OUTCOMES:
The alignment of femoral and tibial components after TKA | Within 1 month after operation

CONTACTS AND LOCATIONS:
Overall Officials: Keerati Charoencholvanich, MD, Principal Investigator — Mahidol University

REFERENCES:
- [Derived] Chareancholvanich K, Narkbunnam R, Pornrattanamaneewong C. A prospective randomised controlled study of patient-specific cutting guides compared with conventional instrumentation in total knee replacement. Bone Joint J. 2013 Mar;95-B(3):354-9. doi: 10.1302/0301-620X.95B3.29903. PMID 23450020